CLINICAL TRIAL: NCT03344627
Title: Clinical Outcome Study of High-dose Meropenem in Sepsis and Septic Shock Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Tospon Lertwattanachai, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID07-60-19
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Sepsis; Septic Shock; Critical Illness; Carbapenem; Pharmacokinetic; Pharmacodynamic; Clinical Outcome; Organ Failure, Multiple; Morality
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness; Multiple Organ Failure | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meropenem standard dose (Active Comparator): Meropenem 1 g every 8 hours
  Interventions: Drug: Meropenem standard dose
- Meropenem high dose (Active Comparator): Meropenem 2 g every 8 hours
  Interventions: Drug: Meropenem high dose

INTERVENTIONS:
Drug: Meropenem standard dose — * Empirical with 1 g meropenem intravenous infusion in 30 minutes then 1 g intravenous infusion in 3 hours every 8 hours.
  * Dosage is adjusted in case of renal dysfunction. Duration of therapy is varied regarding source(s) of infection.
  Arms: Meropenem standard dose
Drug: Meropenem high dose — * Empirical with 2 g meropenem intravenous infusion in 30 minutes then 2 g intravenous infusion in 3 hours every 8 hours.
  * Dosage is adjusted in case of renal dysfunction. Duration of therapy is varied regarding source(s) of infection
  Arms: Meropenem high dose

SUMMARY:
Sepsis and septic shock patients are considered to have a high risk of complications and death. Appropriate antimicrobial therapy plays an important role in determining outcomes in septic patients. However, pathophysiologic changes associated with critical illness have an impact on pharmacokinetics of antimicrobials. In addition, increasing bacterial resistance is also a growing concern, especially in intensive care units., Consequently, standard antimicrobial dose may not be sufficient to achieve pharmacokinetic/pharmacodynamic target in sepsis and septic shock patients. The purpose of this study is to compare a therapy between meropenem standard dose and meropenem high dose in the treatment of sepsis and septic shock

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) with sepsis and/or septic shock according to SEPSIS-3 criteria and receive meropenem within 1 hour after diagnosis
* Informed consent signed by patient or their legally authorized representative

Exclusion Criteria:

* Subjects with infective endocarditis
* Subjects with central nervous system infection
* Subjects who requires surgical condition within 72 hours after randomization
* Subjects on extracorporeal membrane oxygenation (ECMO) within 3 days after randomization
* Subjects with active seizure
* History of receiving meropenem within 1 week prior to randomization
* Pregnancy women and lactation
* Known allergy to meropenem
* Not complete a 72-hour course of empirical meropenem treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
SOFA score change | Change from Baseline SOFA score at day 4
  The Sequential organ failure assessment (SOFA) score describe the time course of multiple organ dysfunction.
  The SOFA score is composed of scores for six organ systems (respiratory, cardiovascular, neurological, hepatic, renal and coagulation).
  The function of six organ systems is scored from 0 (no organ dysfunction) to 4 (severe organ dysfunction), and the individual organ scores are then summed to a total score between 0 and 24.
  Primary outcome is assessing change between SOFA score at baseline and SOFA score at day 4 after treatment by meropenem

SECONDARY OUTCOMES:
Mortality | 14 and 28 days
  In hospital mortality
Clinical cure | Day 3, 5, 7, 10 and 14
  Composite of:
  1. Persistent fever and/or
  2. Stable or increased white blood cell count
Microbiological cure | Day 3, 5, 7, 10 and 14
  Elimination of the study entry pathogen within 14 days after received meropenem
  * Bacteremia: no growth in blood cultures
  * Intra-abdominal infection: no growth in blood cultures
  * UTI: uropathogen growth of less than 10^4 CFU/mL in women or less than 10^3 CFU/mL in men
  * HAP/VAP: pathogen in sputum culture growth of less than 10^3 CFU/mL
  * SSTI: no growth in blood cultures
Duration of vasopressor agents | 14 and 28 days
  Time interval (day) from time of vasopressor agents initiation to time to vasopressor agents discontinuation
Duration of mechanical ventilator | 14 and 28 days
  Time interval (day) of mechanical ventilator
Length of ICU stay | 14 and 28 days
  Time interval (day) from ICU admission (after randomization) to ICU discharge
Length of hospital stay | 14 and 28 days
  Time interval (day) from hospital admission (after randomization) to hospital discharge
%T > MIC | Day 1
  % time of meropenem concentration above MIC

CONTACTS AND LOCATIONS:
Overall Officials: Tospon Lertwattanachai, B.sc.(Pharm), Principal Investigator — Faculty of Pharmacy, Mahidol University
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Background] Jaruratanasirikul S, Thengyai S, Wongpoowarak W, Wattanavijitkul T, Tangkitwanitjaroen K, Sukarnjanaset W, Jullangkoon M, Samaeng M. Population pharmacokinetics and Monte Carlo dosing simulations of meropenem during the early phase of severe sepsis and septic shock in critically ill patients in intensive care units. Antimicrob Agents Chemother. 2015;59(6):2995-3001. doi: 10.1128/AAC.04166-14. Epub 2015 Mar 9. PMID 25753628
- [Background] Roberts JA, Kumar A, Lipman J. Right Dose, Right Now: Customized Drug Dosing in the Critically Ill. Crit Care Med. 2017 Feb;45(2):331-336. doi: 10.1097/CCM.0000000000002210. PMID 28098629
- [Background] Suwantarat N, Carroll KC. Epidemiology and molecular characterization of multidrug-resistant Gram-negative bacteria in Southeast Asia. Antimicrob Resist Infect Control. 2016 May 4;5:15. doi: 10.1186/s13756-016-0115-6. eCollection 2016. PMID 27148448
- [Background] Blot SI, Pea F, Lipman J. The effect of pathophysiology on pharmacokinetics in the critically ill patient--concepts appraised by the example of antimicrobial agents. Adv Drug Deliv Rev. 2014 Nov 20;77:3-11. doi: 10.1016/j.addr.2014.07.006. Epub 2014 Jul 15. PMID 25038549
- [Background] Marquet K, Liesenborgs A, Bergs J, Vleugels A, Claes N. Incidence and outcome of inappropriate in-hospital empiric antibiotics for severe infection: a systematic review and meta-analysis. Crit Care. 2015 Feb 16;19(1):63. doi: 10.1186/s13054-015-0795-y. PMID 25888181
- [Background] Mouton JW, van den Anker JN. Meropenem clinical pharmacokinetics. Clin Pharmacokinet. 1995 Apr;28(4):275-86. doi: 10.2165/00003088-199528040-00002. PMID 7648757
- [Background] de Grooth HJ, Geenen IL, Girbes AR, Vincent JL, Parienti JJ, Oudemans-van Straaten HM. SOFA and mortality endpoints in randomized controlled trials: a systematic review and meta-regression analysis. Crit Care. 2017 Feb 24;21(1):38. doi: 10.1186/s13054-017-1609-1. PMID 28231816
- [Derived] Lertwattanachai T, Montakantikul P, Tangsujaritvijit V, Sanguanwit P, Sueajai J, Auparakkitanon S, Dilokpattanamongkol P. Clinical outcomes of empirical high-dose meropenem in critically ill patients with sepsis and septic shock: a randomized controlled trial. J Intensive Care. 2020 Apr 15;8:26. doi: 10.1186/s40560-020-00442-7. eCollection 2020. PMID 32318268